CLINICAL TRIAL: NCT02012179
Title: The Long Term Effects of Dietary Sodium Restriction on Clinical Outcomes in Patients With Heart Failure
Brief Title: SODIUM-HF: Study of Dietary Intervention Under 100 MMOL in Heart Failure
Acronym: SODIUM-HF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MOP130275
Record Dates: First submitted 2013-12-10; First posted 2013-12-16 (Estimated); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Heart Failure
Keywords: Diet; Dietary sodium reduction; Salt restriction; Nutrition
MeSH Terms: conditions — Heart Failure | interventions — Diet, Sodium-Restricted

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low sodium diet (Experimental): Low sodium diet (65 mmol or 1500 mg/day)
  Interventions: Other: Low sodium diet
- Usual Care (No Intervention): General advice to limit dietary sodium as it is provided during routine clinic practice

INTERVENTIONS:
Other: Low sodium diet — Low sodium diet (65 mmol or 1500 mg/day)
  Arms: Low sodium diet

SUMMARY:
SODIUM-HF is a multicenter clinical trial in ambulatory patients with chronic HF to evaluate the efficacy of a low sodium containing diet on a composite clinical outcome composed of of all-cause mortality, cardiovascular hospitalizations and cardiovascular emergency department visits. The hypothesis of this study is that patients following a low-sodium containing diet will have fewer clinical events (fewer hospital readmissions or emergency department visits, longer survival) than those randomized to Usual Care.

ELIGIBILITY:
Inclusion Criteria:

* Patients recruited if they are 18+ years or older, with confirmed diagnosis of HF (both reduced and preserved systolic function are eligible), NYHA class II-III, and willing to sign informed consent.

Exclusion Criteria:

Subjects will be excluded if:

* Average dietary intake of <1500 mg/ day by a quantitative or semi-quantitative method
* Serum sodium <130mmol/L
* Renal failure (glomerular filtration rate <30 mL/min)
* Hepatic failure
* Uncontrolled thyroid disorder
* Cardiac device (ICD or CRT) or revascularization procedure (PCI or CABG) in previous month or planned in next 3 months
* Hospitalization due to cardiovascular causes in previous 1 month
* Uncontrolled atrial fibrillation (resting heart rate >90 bpm)
* Active malignancy
* Moderate-severe dementia
* Enrolled in another interventional research study
* Patients will be excluded, if in the opinion of the investigator, another condition exists that would preclude dietary compliance or compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 806 (Actual)
Dates: Start 2014-03-24 (Actual); Primary Completion 2022-09 (Actual); Study Completion 2023-01 (Actual)

PRIMARY OUTCOMES:
Composite Clinical Outcomes | 12 months
  All-cause mortality, cardiovascular hospitalizations or cardiovascular emergency department visits

SECONDARY OUTCOMES:
Exercise capacity | 12 months
  Change in exercise capacity as measured by the 6-minute walk test (6MWT)
NYHA functional class | 12 months
  Change in NYHA class treated as a categorical variable
Quality of life (KCCQ) | 12 months
  Change in quality of life assessed by the KCCQ

CONTACTS AND LOCATIONS:
Overall Officials: Justin Ezekowitz, MBBCh, Principal Investigator — University of Alberta
Locations (26):
- Australia (3):
  - The Prince Charles Hospital, Chermside
  - St. Vincent's Hospital Sydney, Darlinghurst
  - Metro North Hospital and Health Service, Herston
- Canada (17):
  - University of Calgary / Foothills Medical Centre, Calgary, Alberta
  - St. Mary's Hospital, Camrose, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Red Deer Regional Hospital, Red Deer, Alberta
  - Private Cardiology Practice, Delta, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - St. Boniface Hospital, Winnipeg, Manitoba
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Brampton Research Associates, Brampton, Ontario
  - Hamilton Health Sciences, Hamilton, Ontario
  - Southlake Regional Health Centre, Newmarket, Ontario
  - Curans Heart Centre, Thunder Bay, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Prairie Vascular Research Inc., Regina, Saskatchewan
  - Royal University Hospital, Saskatoon, Saskatchewan
- Chile (2):
  - Hospital Base Osorno, Osorno
  - Centro de estudios cardiologicas y de Medicine Interna Ltda (Centre for Cardiology and Internal Medicine Studies), Temuco
- Unidad de Investigación en Epidemiología Clínica Hospital General Regional No. 1, IMSS, Mexico City, Mexico
- New Zealand (3):
  - Middlemore Clinical Trials, Auckland
  - University of Auckland, Auckland
  - Christchurch Heart Institute / University of Otago, Christchurch

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ezekowitz JA, Colin-Ramirez E, Ross H, Escobedo J, Macdonald P, Troughton R, Saldarriaga C, Alemayehu W, McAlister FA, Arcand J, Atherton J, Doughty R, Gupta M, Howlett J, Jaffer S, Lavoie A, Lund M, Marwick T, McKelvie R, Moe G, Pandey AS, Porepa L, Rajda M, Rheault H, Singh J, Toma M, Virani S, Zieroth S; SODIUM-HF Investigators. Reduction of dietary sodium to less than 100 mmol in heart failure (SODIUM-HF): an international, open-label, randomised, controlled trial. Lancet. 2022 Apr 9;399(10333):1391-1400. doi: 10.1016/S0140-6736(22)00369-5. Epub 2022 Apr 2. PMID 35381194
- [Derived] Colin-Ramirez E, Ezekowitz JA; SODIUM-HF investigators. Rationale and design of the Study of Dietary Intervention Under 100 MMOL in Heart Failure (SODIUM-HF). Am Heart J. 2018 Nov;205:87-96. doi: 10.1016/j.ahj.2018.08.005. Epub 2018 Aug 16. PMID 30205241